CLINICAL TRIAL: NCT01974804
Title: Assessment of Early Treatment Response by Diffusion and Perfusion MRI in Patients With Brain Metastasis
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 13-094
Record Dates: First submitted 2013-10-28; First posted 2013-11-04 (Estimated); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Brain Cancer
Keywords: MRI; Brain metastases; 13-094
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pts having an MRI: Patients will undergo a 20 minute pretreatment MRI scan and a 30 minute post treatment MRI scan with contrast agent administration. Ten patients with brain metastasis will be recruited in the study. All the patients will be undergoing SRS (Stereotactic Radiosurgery). Patients will have 1 pretreatment evaluation and 2 post treatment evaluations [1-72 hours post treatment and 8 weeks (+/- 2 weeks) post treatment] for early response. Patients are to be administered contrast prior to obtaining MRI scans. These research scans are estimated to take 20 minutes of scan time (+/- 10 minutes), which includes patient set up and conducting the research sequences..
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI

SUMMARY:
Magnetic resonance imaging (MRI) is a diagnostic study that makes pictures of organs of the body using magnetic field and radio frequency pulses that can not be felt. The purpose of this study is to determine if new imaging methods can help tumor evaluation in the brain. The extra images will be obtained using diffusion and perfusion MRI techniques to assess early treatment response in patients with brain metastasis, and will be compared to methods currently being used.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and over.
* Patients/Subjects able to give informed consent
* Patients/Subjects whose weight does not exceed 275 lbs.
* Patient with metastatic brain tumors greater than or equal to 1.0 cm that will be treated with stereotactic radiosurgery and scheduled for an MRI scan as part of their routine care

Exclusion Criteria:

* Patients who are unwilling or unable to undergo MRI including patients with contra-indications to MRI such as the presence of cardiac pacemakers or non-compatible intracranial vascular clips.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The protocol investigators on the study will identify potential research participants from those patients who are scheduled for MRI examination as part of their routine clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-10-25 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
feasibility of diffusion and perfusion magnetic resonance imaging (MRI) | 1 year
  This is a technology assessment protocol for response to treatment. The study is designed to assess the utility of the technology using a limited number of participants. We will assess whether the MR parameters are predictive markers of early response.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Beal, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/